CLINICAL TRIAL: NCT04628286
Title: Effects of Myofascial Induction Technique in Stabilometry Plantar Fascia Compared to a Placebo Laser
Brief Title: Myofascial Induction Effects on Stabilometry Versus Sham Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Head of Podiatry, Principal Investigator, and Physiotherapist, Mayuben Private Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2111201814518 C
Record Dates: First submitted 2020-11-07; First posted 2020-11-13 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Foot Diseases; Myofascial Pain
MeSH Terms: conditions — Foot Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Laser (Placebo Comparator): Placebo laser application in plantar fascia
  Interventions: Other: Sham Laser
- Experimental group Myofascial Induction (Experimental): Myofascial Induction technique application in plantar fascia
  Interventions: Other: Myofascial Induction

INTERVENTIONS:
Other: Sham Laser — Sham Laser in plantar fascia
  Arms: Sham Laser
Other: Myofascial Induction — Myofascial Induction in plantar fascia
  Arms: Experimental group Myofascial Induction

SUMMARY:
The objective is to determine the effectiveness of myofascial induction effects on stabilometric variables. Forty healthy subjects will be recruited for a single blind clinical trial. All subjects will be randomly distributed into two different groups: control group (simulated laser) and experimental group (myofascial induction). Result measurements will be performed in the center of the pressure area (stabilometry) using a validated platform. Two trials will be recorded for each condition (eyes closed and eyes open)

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals without pain.

Exclusion Criteria:

* Previous lower extremities surgery
* History of lower extremities injury with residual symptoms within the last year
* Evidence of a leg-length discrepancy of more than 1 cm
* Evidence of balance deficits

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Stabilometry variable eyes open before Sham Laser or Myofascial Induction | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º from the midline. Stabilometric variables measure the displacement of the center of pressures in X (in millimeters) with the eyes open.
Stabilometry variables eyes open before Sham Laser or Myofascial indution | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned 30º from the midline. The stabilometry variables measure the displacement of the center of pressures in Y (in millimeters) with the eyes open.
Stabilometry variables eyes open before Sham Laser or Myofascial indution | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of Pressure (COP) area (in millimeters²) with eyes open.
Stabilometry variables eyes open before Sham Laser or Myofascial indution | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned 30º from the midline. Stabilometric variables measure the center of pressure and the velocity displacement of the anteroposterior direction (a-p) (in millimeters / second).
Stabilometry variables eyes open before Sham Laser or Myofascial indution | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned 30º from the midline. Stabilometric variables measure center of pressure, velocity, and lateral-lateral (lat-lat) direction displacement (in millimeters / second).
Stabilometry variables eyes closed before Sham Laser or Myofascial indution | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º from the midline. The stabilometric variables measure the displacement of the center of pressures in X (in millimeters) with the eyes closed.
Stabilometry variables eyes closed before Sham Laser or Myofascial indution | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned 30º from the midline. The stabilometry variables measure the displacement of the center of pressures in Y (in millimeters) with the eyes closed.
Stabilometry variables eyes closed before Sham Laser or Myofascial indution | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned 30º from the midline. The stabilometry variables measure the displacement of the area of the center of pressure (COP) (in millimeters²) with the eyes closed.
Stabilometry variables eyes closed before Sham Laser or Myofascial indution | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned 30º from the midline. Stabilometric variables measure the center of pressure and the velocity displacement of the anteroposterior direction (a-p) (in millimeters / second).
Stabilometry variables eyes closed before Sham Laser or Myofascial indution | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned 30º from the midline. Stabilometric variables measure center of pressure, velocity, and lateral-lateral (lat-lat) direction displacement (in millimeters / second).
Stabilometry variables eyes open after Sham Laser or Myofascial Induction | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned 30º from the midline. Stabilometric variables measure the displacement of the center of pressures in X (in millimeters) with the eyes open.
Stabilometry variables eyes open after Sham Laser or Myofascial Induction | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned 30º from the midline. The stabilometry variables measure the displacement of the center of pressures in Y (in millimeters) with the eyes open.
Stabilometry variables eyes open after Sham Laser or Myofascial Induction | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º from the midline. Stabilometric variables measure the displacement of the area of the center of pressure (COP) (in millimeters²) with the eyes open.
Stabilometry variables eyes open after Sham Laser or Myofascial Induction | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned 30º from the midline. Stabilometric variables measure the center of pressure and the velocity displacement of the anteroposterior direction (a-p) (in millimeters / second).
Stabilometry variables eyes open after Sham Laser or Myofascial Induction | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned 30º from the midline. Stabilometric variables measure center of pressure, velocity, and lateral-lateral (lat-lat) direction displacement (in millimeters / second).
Stabilometry variables eyes closed after Sham Laser or Myofascial Induction | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned 30º from the midline. The stabilometric variables measure the displacement of the center of pressures in X (in millimeters) with the eyes closed.
Stabilometry variables eyes closed after Sham Laser or Myofascial Induction | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º from the midline. The stabilometry variables measure the displacement of the center of pressures in Y (in millimeters) with the eyes closed.
Stabilometry variables eyes closed after Sham Laser or Myofascial Induction | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned 30º from the midline. Stabilometric variables measure the displacement of the area of the center of pressure (COP) (in millimeters²) with the eyes closed.
Stabilometry variables eyes closed after Sham Laser or Myofascial Induction | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º from the midline. Stabilometry variables measure the center of pressure, the velocity displacement from the anteroposterior direction (a-p) (in millimeters / second).
Stabilometry variables eyes closed after Sham Laser or Myofascial Induction | Through study completion, an average of 1 week
  tabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned 30º from the midline. Stabilometric variables measure center of pressure, velocity, and lateral-lateral (lat-lat) direction displacement (in millimeters / second).

CONTACTS AND LOCATIONS:
Locations (1):
- Mayuben Clinic, San Sebastián de los Reyes, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided